CLINICAL TRIAL: NCT01749969
Title: A Phase 1b Study of SAR650984 (Anti-CD38 mAb) in Combination With Lenalidomide and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: SAR650984 (Isatuximab), Lenalidomide, and Dexamethasone in Combination in RRMM Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD11863; U1111-1119-3107 (Other: UTN)
Record Dates: First submitted 2012-12-10; First posted 2012-12-17 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR650984 (isatuximab) (Experimental): SAR650984 (isatuximab) (escalating dose) plus lenalidomide 25 mg on Days 1 to 21 plus dexamethasone 40 mg on Days 1, 8, 15, 22 in 28-day cycles for all cohorts up to disease progression.
  For Q2W cohorts: SAR650984 (isatuximab) on Days 1 and 15 of every cycle. For QW/Q2W cohorts: SAR650984 (isatuximab) on Days 1, 8, 15, and 22 of first cycle and Days 1 and 15 of every subsequent cycle.
  Interventions: Drug: isatuximab SAR650984; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: isatuximab SAR650984 — Pharmaceutical form:solution Route of administration: intravenous
  Other Names: Sarclisa
Drug: lenalidomide — Pharmaceutical form:capsules Route of administration: oral
  Other Names: Revlimid
Drug: dexamethasone — Pharmaceutical form:solution or tablet Route of administration: intravenous or oral

SUMMARY:
Primary Objectives:

* To determine the maximum tolerated dose of SAR650984 (isatuximab) with lenalidomide and dexamethasone (LD) in patients with relapsed or refractory multiple myeloma.
* Expansion Phase Only: To further evaluate preliminary evidence of antitumor activity (objective response rate [ORR]) of SAR650984 (isatuximab) in combination with LD using International Myeloma Working Group (IMWG) criteria.

Secondary Objectives:

* To evaluate the safety, including immunogenicity, of SAR650984 (isatuximab) in combination with LD in relapsed or refractory multiple myeloma. The severity, frequency and incidence of all toxicities will be assessed.
* To evaluate the pharmacokinetics (PK) of SAR650984 (isatuximab) when administered in combination with LD and the PK of lenalidomide in combination with SAR650984 and dexamethasone.
* To assess the relationship between clinical (adverse event [AE] and/or tumor response) effects and pharmacologic parameters (PK/pharmacodynamics), and/or biologic (correlative laboratory) results.
* For the dose expansion phase, estimate the activity (ORR) using IMWG defined response criteria of SAR650984 (isatuximab) plus LD.
* To describe progression-free survival (PFS) in patients treated with this combination.

DETAILED DESCRIPTION:
The study duration for an individual patient will include a screening period for inclusion of up to 21 days, and at least 4 weeks of treatment in the absence of severe adverse reaction, dose limiting toxicity or disease progression plus up to 60 days post-treatment follow up. The treatment period may continue until disease progression, intolerable toxicity, or Investigator, sponsor, or patient decision to discontinue therapy. After study treatment discontinuation, an end of treatment (EOT) visit will be done at 30 days to assess safety, and at 30 and 60 days for anti-drug antibody (ADA) and PK. If the ADA is positive or inconclusive at day 60, then PK and ADA will be repeated every 30 days until ADA is negative. Patients who discontinue treatment for reasons other than progression of disease will be followed monthly until progression, initiation of subsequent therapy, or until the primary analysis cutoff date, whichever comes first.

ELIGIBILITY:
Inclusion criteria:

Male or female patients age 18 years or older. Diagnosis of multiple myeloma and documentation of at least 2 prior therapies (induction therapy, autologous stem cell transplant, consolidation and maintenance therapy is considered one prior therapy); there is no maximum number of prior regimens and prior bone marrow transplant is acceptable.

Confirmed evidence of disease progression from immediately prior MM therapy or refractory to the immediately prior therapy.

Patients may have received prior immunomodulatory drugs (IMiDs®) (eg, lenalidomide or thalidomide).

Patients with measurable disease. Patients with a Karnofsky ≥60% performance status. Females of childbearing potential (FCBP). Voluntary written informed consent before performance of any study-related procedure not part of routine medical care with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Able to take aspirin daily as prophylactic anti-coagulation therapy (patients intolerant to aspirin may use warfarin, low molecular weight heparin or equivalent anti-platelet therapy).

Adequate organ function.

Exclusion criteria:

Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy.

Prior anti-cancer therapy (chemotherapy, targeted agents, radiotherapy, and immunotherapy) within 21 days except for alkylating agents (eg, melphalan) where 28 days will be required or participated in another clinical trial during the past 30 days.

History of significant cardiovascular disease within the past 6 months, unless the disease is well-controlled.

Prior autologous stem cell transplant within 12 weeks of the first dose of study treatment and/or prior allogeneic transplant within 1 year or has evidence of active graft-versus-host disease (GVHD) requiring >10 mg prednisone daily.

Daily requirement for corticosteroids (>10 mg prednisone qd for 7 consecutive days) (except for inhalation corticosteroids and patients being treated for adrenal insufficiency/replacement therapy).

Evidence of mucosal or internal bleeding. Prior radiation therapy or major surgical procedure within 4 weeks of the first dose of study treatment.

Known active infection requiring parenteral or oral anti-infective treatment. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation.

Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient.

Hypersensitivity to any of the components of study therapy that is not amenable to premedication with steroids and H2 blockers.

Known human immunodeficiency virus (HIV) or active hepatitis B or C viral infection.

Neuropathy ≥ Grade 3 or painful neuropathy ≥ Grade 2. Gastro-intestinal abnormalities, including bowel obstruction, inability to take oral medication, requirement for intravenous (IV) alimentation, active peptic ulcer or prior surgical procedures or bowel resection affecting absorption.

Pregnancy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events when treated with SAR650984 (isatuximab) in combination with LD | Up to 30 days for patients experiencing progressive disease and continuously while patients are on treatment

SECONDARY OUTCOMES:
Preliminary assessment of overall response rate | 9 months from the last investigational medicinal product (IMP)/non-IMP (NIMP) administration
Preliminary assessment of progression-free survival (PFS) | Up to disease progression
Assessment of PK parameters - maximum concentration (Cmax) | Up to disease progression plus 60 days
Assessment of PK parameters - time to reach Cmax (Tmax) | Up to disease progression plus 60 days
Assessment of PK parameters - concentration observed at end of infusion (Ceoi) | Up to disease progression plus 60 days
Assessment of PK parameters - area under the plasma concentration versus time curve over the dosing interval (AUCtau) | Up to disease progression plus 60 days
Assessment of PK parameters - plasma concentration observed just before treatment administration during repeated dosing (Ctrough) | Up to disease progression plus 60 days
Number of CD38 receptors occupied by SAR650984 (isatuximab) | Up to disease progression plus 60 days
CD38 receptor density | Up to disease progression plus 60 days
Immunogenicity: Number of anti-SAR650984 (isatuximab) antibodies in response to SAR650984 (isatuximab) | Up to disease progression plus 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (5):
  - Investigational Site Number 840004, San Francisco, California
  - Investigational Site Number 840001, Tampa, Florida
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840005, New York, New York
  - Investigational Site Number 840003, Columbus, Ohio

REFERENCES:
- [Derived] Sun H, Martin TG, Marra J, Kong D, Keats J, Mace S, Chiron M, Wolf JL, Venstrom JM, Rajalingam R. Individualized genetic makeup that controls natural killer cell function influences the efficacy of isatuximab immunotherapy in patients with multiple myeloma. J Immunother Cancer. 2021 Jul;9(7):e002958. doi: 10.1136/jitc-2021-002958. PMID 34272304
- [Derived] Martin T, Baz R, Benson DM, Lendvai N, Wolf J, Munster P, Lesokhin AM, Wack C, Charpentier E, Campana F, Vij R. A phase 1b study of isatuximab plus lenalidomide and dexamethasone for relapsed/refractory multiple myeloma. Blood. 2017 Jun 22;129(25):3294-3303. doi: 10.1182/blood-2016-09-740787. Epub 2017 May 8. PMID 28483761